CLINICAL TRIAL: NCT04404595
Title: Open-label, Multicenter, Phase 1b/2 Clinical Trial to Evaluate the Safety and Efficacy of Autologous Anti-claudin 18.2 Chimeric Antigen Receptor T-cell Therapy in Subjects with Advanced Gastric, Pancreatic, or Other Specified Digestive System Cancers
Brief Title: Claudin18.2 CAR-T (CT041) in Patients with Gastric, Pancreatic Cancer, or Other Specified Digestive Cancers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT041-ST-02
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer; Pancreatic Cancer
Keywords: CAR-T
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation and expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- anti-claudin18.2 chimeric antigen receptor T-cell therapy (Experimental): Phase 1b will include two parts, dose escalation phase (Cohort A) followed by a dose expansion phase (Cohort B). Phase 2 (Cohort C) will evaluate the chosen dose in patients with advanced gastric cancer.
  Interventions: Biological: CT041

INTERVENTIONS:
Biological: CT041 — treatment with anti-claudin18.2 chimeric antigen receptor T-cell infusion

SUMMARY:
A Phase 1b/2, open label, multi-center, clinical study of Chimeric Antigen Receptor T Cells (CAR-T) targeting claudin18.2 in patients with advanced gastric, pancreatic or other specified digestive system cancers

DETAILED DESCRIPTION:
This is an open label, multi-center, Phase 1b/2 clinical trial to evaluate the safety and efficacy of autologous claudin18.2 chimeric antigen receptor T-cell therapy in patients with advanced gastric, pancreatic or other specified digestive system cancers.

Following consent, patients must have tumor tissue evaluated by CLDN18.2 IHC assay. Patients meeting all eligibility criteria will undergo a leukapheresis procedure to collect autologous mononuclear cells for manufacture of investigational drug product (CT041). Following manufacture of the drug product, subjects will receive preconditioning prior to CT041 infusion. All subjects will be asked to continue to undergo long-term gene safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for screening for potential inclusion in the study (* indicates inclusion criteria at Baseline (for subjects to be eligible for preconditioning)):

1. Voluntarily signed the ICF;
2. Age ≥ 18 and < 76 years with pathologically/histologically confirmed diagnosis of adenocarcinoma of the stomach or gastroesophageal junction, referred to collectively as STAD, or pancreatic adenocarcinoma (PAAD);or biliary tract cancers (BTCs, including intrahepatic/extrahepatic cholangiocarcinoma and gallbladder cancer but not ampullary carcinoma);
3. Must have CLDN18.2-positive tumor expression as determined by the CLDN18.2 IHC assay;
4. Estimated life expectancy > 4 months*;
5. Failed or been intolerant of prior lines of systemic therapy:

   1. For screening:

      * Leukapheresis can be performed for subjects with STAD who have progressed or were intolerant of at least 1 prior line of systemic therapy, or,
      * Leukapheresis can be performed for subjects with PAAD who are receiving first-line treatment, or,
      * Leukapheresis can be performed for subjects with BTC who are receiving first-line treatment.
   2. Baseline*:

      * Subjects with STAD who have progressed or were intolerant of at least 2 prior lines of systemic therapy, or,
      * Subjects with PAAD who have progressed or were intolerant of at least 1 prior line of systemic therapy, or,
      * Subjects with BTC who have progressed or were intolerant of at least 1 prior line of systemic therapy. For subjects with CCA with who has FGFR2 fusions or rearrangements, or IDH1-mutant must have received FDA-approved target therapies.
6. At least 1 measurable lesion per RECIST 1.1*;
7. ECOG performance status of 0 or 1*;
8. Sufficient venous access for leukapheresis collection and no other contraindications to leukapheresis;
9. Patients should have adequate CBC counts, renal and hepatic functions*;
10. Women of childbearing age must undergo a serum pregnancy test with negative results before screening and infusion and be willing to use effective and reliable method of contraception*;
11. Men must be willing to use effective and reliable method of contraception for at least 12-months after T-cell infusion*;
12. Sufficient nutritional status.

Exclusion Criteria for screening (* indicates exclusion criteria for baseline as well):

1. Pregnant or lactating women*;
2. HIV, active hepatitis C virus (HCV), active hepatitis B virus (HBV), or active syphilis infection;
3. Any active infection requiring systemic treatment*;
4. AEs from previous treatment that have not recovered*;
5. Patients who have clinically significant thyroid dysfunction;
6. Patients allergic to any drugs of the preconditioning regimen, tocilizumab, dimethyl sulfoxide (DMSO), or CT041 CAR-CLDN18.2 T-cell;
7. Patients who have received:

   1. prior cellular therapy such as (CAR T, TCR, tumor-infiltrating lymphocytes) within one year.
   2. organ transplantation.
   3. previous anti-claudin18.2 CAR T-cell therapy, mRNA-based cancer immunotherapy, or bispecific T cell engager.
8. Untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression;
9. Patients with heavy tumor burdens;
10. Unstable/active ulcer, anastomotic recurrence with full-thickness tumor infiltration or tumor involving any major vessels, digestive tract bleeding, or recent digestive surgery that may have increased risk of bleeding*;
11. Patients who have a history of esophageal or gastric resection plus current evidence of locally recurrent tumor that involves any major blood vessels or that has evidence of recent bleeding or perforation*;
12. Patients requiring anticoagulant therapy such as warfarin or heparin;
13. Patients requiring long-term antiplatelet therapy;
14. Use of prednisone >/= 10mg daily or other equivalent steroids within 14 days before leukapheresis or preconditioning*;
15. Anticancer treatment within approximately 2 weeks prior to leukapheresis or preconditioning*;
16. Major surgery less than 1 week prior to leukapheresis or 3 weeks prior to preconditioning*;
17. Patients who have clinically significant cardiac conditions that researchers believe that participating in this clinical trial may endanger the health of the patients*;
18. Inadequate pulmonary function*;
19. Patients known to have active autoimmune diseases;
20. Patients with second malignancies;
21. Patients have significant neurologic disorders;
22. Patients are unable or unwilling to comply with the requirements of clinical trial.

    Additional exclusion criteria solely for baseline (prior to conditioning regimen):
23. Fever > 38.0°C;
24. Active illness or existing toxicity that would place the subject at undue risk;
25. Abrupt deterioration of clinical status or condition;
26. Subjects who have received a live attenuated vaccine 4 weeks before preconditioning.

Inclusion Criteria Before Infusion: There are no inclusion criteria at this timepoint.

Exclusion Criteria Before Infusion:

1. Patients who have clinically significant cardiac conditions that researchers believe that participating in this clinical trial may endanger the health of the patients;
2. Inadequate pulmonary function;
3. Active infection requiring systemic therapy or causing fever within 7 days prior to investigational infusion;
4. Active illness or toxicity that would place the subject at undue risk;
5. Abrupt deterioration of clinical status or condition;
6. New or worsening Grade ≥ 3 non-hematologic toxicities.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1b (Cohort A): Evaluate the safety and tolerability of CAR-CLDN18.2 T-cell therapy (CT041) in subjects with specified advanced digestive system cancers (STAD, PAAD, or BTC). | up to year 15
  Incidence of adverse events (AEs), AEs of special interest (cytokine release syndrome [CRS], neurotoxicity, secondary malignancy), serious adverse events (SAEs).
Phase 1b (Cohort A): Identify the recommended Phase 2 dose (RP2D) of CT041 therapy in subjects with advanced STAD, PAAD, or BTC. | day 0 - day 28
  Incidence of dose-limiting toxicities (DLTs)
Phase 1b (Cohort A): Identify the maximum tolerated dose (MTD) or maximum administered dose (MAD) of CT041 therapy in subjects with STAD, PAAD, or BTC. | day 0 - day 28
  The highest dose below the dose where the escalation was stopped when the frequency or severity of DLTs exceeds predefined safety criteria.
Phase 1b (Cohort B): Determine the efficacy of CT041 by ORR in subjects with advanced STAD, PAAD, or BTC. | up to year 15
  Objective response rate by IRC assessment (RECIST v1.1)
Phase 2 (Cohort C): Determine the efficacy of CT041 by ORR in subjects with advanced STAD treated at the RP2D. | up to year 15
  Objective response rate by IRC assessment (RECIST v1.1)

SECONDARY OUTCOMES:
Phase 1b/2: Objective Response Rate (ORR) per investigator assessment | up to year 15
  Rate of subjects experiencing an objective response (a binary variable indicating whether each subject experienced a ≥ partial response [PR] by Response Evaluation Criteria in Solid Tumors, version 1.1 [RECIST 1.1]), as determined by investigator assessment.
Phase 1b (Cohort A): Duration of Response | up to year 15
  Duration of time from first response to progression of disease as determined by investigator
Phase 1b (Cohort A): Time to Progression | up to year 15
  Duration of time in months from the date of CT041 infusion until disease progression, excluding deaths as determined by investigator.
Phase 1b (Cohort A): Disease Control Rate | up to year 15
  The incidence of a BOR of CR, PR, or SD based on investigator assessments using RECIST 1.1 criteria.
Phase 1b (Cohort A): Progression free survival | up to year 15
  The time in months from the date of CT041 infusion to the earliest date of disease progression or death due to any cause as determined by investigator.
Phase 1b (Cohort B): Evaluate the safety and tolerability of CAR-CLDN18.2 T-cell therapy (CT041) in subjects with specified advanced digestive system cancers (STAD, PAAD, or BTC). | up to year 15
  Incidence of adverse events (AEs), AEs of special interest (cytokine release syndrome [CRS], neurotoxicity, secondary malignancy), serious adverse events (SAEs).
Phase 2 (Cohort C): Evaluate the safety and tolerability of CAR-CLDN18.2 T-cell therapy (CT041) in subjects with advanced STAD. | up to year 15
  Incidence of adverse events (AEs), AEs of special interest (cytokine release syndrome [CRS], neurotoxicity, secondary malignancy), serious adverse events (SAEs).
Phase 1b(Cohort B)/2: Duration of Response | up to year 15
  Duration of time from first response to progression of disease as determined by investigator and IRC assessment.
Phase 1b(Cohort B)/2: Time to Progression | up to year 15
  Duration of time in months from the date of CT041 infusion until disease progression, excluding deaths as determined by investigator and IRC assessment.
Phase 1b(Cohort B)/2: Disease Control Rate | up to year 15
  The incidence of a BOR of CR, PR, or SD based on investigator and IRC assessments using RECIST 1.1 criteria.
Phase 1b(Cohort B)/2: Progression free survival | up to year 15
  The time in months from the date of CT041 infusion to the earlier date of disease progression or death due to any cause as determined by investigator and IRC assessment.
Phase 1b/2: Overall survival | up to year 15
  The time in months from the date of CT041 infusion until the date of death by any cause.
Phase 1b/2: Utilization of Hospital Resources | Day 0 to 3 months
  Total days of hospitalization, including ICU days, during & after CT041 infusion as described below:
  * Infusion-related hospital re-admission within 3 months after infusion.
  * The number and percentages of subjects, and the number of hospitalizations due to non-infusion reasons.
  * All-cause re-admission within 3 months after infusion, and from infusion to data cutoff date among those who required rehospitalization
  * Duration of hospitalization in intensive care
Phase 1b(Cohort B)/2: PK and bio-distribution of CT041 | Baseline - month 18
  CAR transgene copy number, peak value, AUC, in vivo persistence.
Phase 1b(Cohort B)/2: Health-related Quality of Life (HRQoL) in STAD patients (Cohorts B & C) | Baseline - month 18
  * Change from baseline in HRQoL as measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30.
  * Change from baseline in HRQoL as measured by EORTC QLQ-OG25.
Phase 1b(Cohort B)/2: CLDN18.2 ICH Assay Performance | Baseline - month 18
  * Association of CLDN18.2 expression level versus tumor response
  * Association of CLDN18.2 expression versus clinical disease characteristics
Phase 1b(Cohort B)/2: Cytokine expression level in blood after CT041 infusion | Baseline - week 20
  Evaluate cytokine expression level in blood after CT041 infusion.
Phase 1b (Cohort B)/2: Anti-CT041 drug antibodies | Baseline - month 12
  Number of subjects with anti-CT041 drug antibodies
Phase 1b (Cohort B)/2: CT041 product characteristics | Baseline - month 18
  Association of CT041 product characteristics with clinical safety/efficacy/PK
Phase 1b (Cohort B)/2: Concordance analysis | up to year 15
  Concordance analysis of ORR of IRC assessment vs investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Harry H Yoon, MD, Principal Investigator — Mayo; Dae Won Kim, MD, Principal Investigator — Moffitt
Locations (16):
- United States (15):
  - City of Hope, Duarte, California
  - University of Southern California, Los Angeles, California
  - UCSD, San Diego, California
  - UCSF, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Karmanos Cancer Center, Detroit, Michigan
  - Mayo Cancer Hospital, Rochester, Minnesota
  - Northwell Cancer Institute, New Hyde Park, New York
  - The Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - TX Oncology-Baylor Charles Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Botta GP, Chao J, Ma H, Hahn M, Sierra G, Jia J, Hendrix AY, Nolte Fong JV, Ween A, Vu P, Miller A, Choi M, Heyman B, Daniels GA, Kaufman D, Jamieson C, Li Z, Cohen E. Metastatic gastric cancer target lesion complete response with Claudin18.2-CAR T cells. J Immunother Cancer. 2024 Feb 5;12(2):e007927. doi: 10.1136/jitc-2023-007927. PMID 38316518